CLINICAL TRIAL: NCT06891703
Title: Phase 1 Study to Evaluate [18F]ACI-15916 as a Potential PET Radioligand for Imaging α-synuclein Deposits in the Brain of Patients With Suspected α-synuclein Pathology Compared With Healthy Volunteers
Brief Title: [18F]ACI-15916 PET in α-synucleinopathies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: AC Immune SA (Industry)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACI-15916-PD-2401; 2024-515664-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease (PD); Multiple System Atrophy (MSA); Dementia With Lewy Bodies (DLB)
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with suspected α-synucleinopathies (Experimental): The study population will be composed of participants with suspected α-synucleinopathies
  Interventions: Other: [18F]ACI-15916
- Healthy volunteers (Active Comparator): The study population will be composed of healthy volunteers
  Interventions: Other: [18F]ACI-15916

INTERVENTIONS:
Other: [18F]ACI-15916 — [18F]ACI-15916 is an intravenously administered radioactive imaging agent being studied as a potential positron emitting radiopharmaceutical for in vivo imaging of α-synuclein deposits.

SUMMARY:
The goal of this clinical trial is to test whether we can reliably and safely measure the accumulation of pathological protein α-synuclein [involved in some diseases such as Parkinson's disease, Lewy body dementia and Multiple System Atrophy (MSA), collectively named α-synucleinopathies] using a new positron emission tomography (PET) tracer called [18F]ACI-15916. Both healthy people and people with (suspected) α-synuclein pathology will participate to this trial.

The main questions it aims to answer are:

* whether [18F]ACI-15916 is safe and well tolerated when injected into participants
* whether [18F]ACI-15916 reliably detects α-synuclein in the brain using PET technique.
* whether there are differences in the amount of this protein between people with diseases related to α-synuclein accumulation in the brain and people without these diseases.

Participants will:

* Visit the clinic to consent to their participation and to ensure they are eligible [physical and neurological examinations, questionnaires, blood and urine tests, ECG and in some cases a MRI and a PET scan with a licensed tracer ([18F]FE-PE2I) to confirm or not the disease].
* Visit the clinic to receive the tracer [18F]ACI-15916 intravenously and be scanned in a PET scanner, during which blood will be collected (and optionally spinal fluid).
* Receive a phone call from the clinic 1 week after the PET scan to report any symptoms and side-effects that they may be having.

Some of the participants may be asked to come again to the clinic for a second PET scan with [18F]ACI-15916, allowing the researchers to determine if the measurements with the first PET scan are stable and reproducible.

Some of the participants will participate in a specific part of the study to evaluate the distribution of the PET ligand in the whole body, with a similar visit schedule.

DETAILED DESCRIPTION:
This is an open-label, first in human (FiH) positron emission tomography (PET) microdose study in patients with suspected α-synuclein pathology and healthy volunteers (HVs) using [18F]ACI-15916 as a novel radioligand. This study will be dedicated to qualification of the ligand [18F]ACI-15916 to measure α-synuclein pathology using PET investigations, including estimation of effective dose and test-retest reliability.

The study consists of four parts in which a total of up to 46 participants may be included:

* Part 1: Up to 5 HVs and up to 5 patients with Parkinson's Disease (PD) will be included.
* Part 2: Up to 30 additional subjects including: HV cases (maximum 10) and patients with α-synucleinopathies such as PD, Multiple System Atrophy (MSA) and Dementia with Lewy Bodies (DLB).
* Part 3: Up to 10 participants from Part 1 and/or Part 2 will have a second PET measurement within one month after their initial PET measurement to evaluate test-retest variability and reproducibility.
* Part 4. Up to 6 HVs (3 female and 3 male) will undergo a whole-body PET-CT examination to estimate the effective dose after one administration of [18F]ACI-15916.

The four study parts can overlap.

The study consists of a screening period of up to 60 days to assess participants' eligibility, a PET scan with [18F]ACI-15916 along with arterial blood sampling, and a safety phone call following the scanning visit. For participants in Part 3, a second PET scan with [18F]ACI-15916 will be performed up to one month after the first scan to evaluate test-retest variability and reproducibility, followed by a new safety phone call. For subjects in Part 4 (dosimetry), no arterial blood sampling will be performed. The total study duration will be up to 10 weeks for Part 1, 2 and 4 participants and up to 14 weeks for Part 3 participants.

ELIGIBILITY:
Inclusion Criteria for all Participants:

1. Subject is able to provide written informed consent, which must be obtained before any assessment is performed.
2. Subjects must be able to understand and be willing to comply with study procedures, restrictions, and requirements.
3. Body mass index is > 18 and < 31 kg/m2 and Bodyweight ≥ 50 kg and ≤ 100 kg.
4. Female participants must not be of childbearing potential or agree to use highly effective methods of contraception.
5. For subjects receiving arterial cannulation, an adequate circulation to the hand for safe placement of arterial line (as determined by Allen's test).

   Additional Inclusion Criteria for Healthy Volunteers:
6. Males and females aged ≥ 20 at the time of signing the informed consent.
7. Normal MRI and DAT PET or SPECT (except for Part 4 participants), as judged by the investigator.
8. The subject is, in the opinion of the investigator, generally healthy based on the assessment of medical history, physical examination, vital signs, ECG, and the results of the hematology, clinical chemistry, urinalysis, serology, and other laboratory tests.
9. No family history of α-synucleinopathy, including PD, or other early-onset neurological disease associated with dementia.
10. No personal history of clinically significant neurologic and/or psychiatric disorders.
11. Have a Montreal Cognitive Assessment (MoCA) score ≥ 26
12. No cognitive impairment as judged by the PI or delegated physician.

    Additional Inclusion Criteria for Participants with α-synucleinopathies:
13. Males and females aged ≥ 40 at the time of signing the informed consent.
14. Subjects diagnosed with any of the following:

    * Idiopathic PD based on MDS criteria
    * PD with genetic risk factor (except some mutations as mentioned in exclusion criteria)
    * Dementia with Lewy bodies (DLB)
    * Diagnosis of possible or probable Multiple System Atrophy (MSA)
15. Evidence of dopamine transporter deficit on DAT PET or SPECT imaging performed either as part of Screening or previously acquired (if not older than 6 months) and of good quality as judged by the investigator.
16. Medications taken for symptomatic treatment of α-synucleinopathy must be maintained on a stable dosage regimen for at least 30 days before the Screening Visit.

Exclusion Criteria for all Participants:

1. Female subjects pregnant, lactating or breastfeeding.
2. Presence of psychiatric symptoms that may interfere with the objectives of the study, as judged by the investigator.
3. Clinically significant concomitant disease or condition within 6 months prior to screening, that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the participant, or compromise the scientific quality of the study.
4. History of brain surgery or any neurosurgical procedures. Subject has received treatment with a drug, antibody or vaccine targeting α-synuclein.
5. Known or suspected drug, alcohol or other abuse, or positive urine drug screen which may interfere with the study objective, as judged by the investigator.
6. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity as judged by the investigator.
7. Subject is involved in the planning and/or conduct of the study (i.e. part of the study team)
8. History of clinically significant cardio-or cerebrovascular, pulmonary, renal, hepatic, neurological, mental or gastrointestinal disorder or any other major disorder that may interfere with the objectives of the study, as judged by the investigator.
9. History of and/or screening brain MRI scan (except for Part 4 subjects) indicative of, clinically significant abnormality including but not limited to prior haemorrhage or infarct or >3 lacunar infarcts, except changes consistent with α-synucleinopathies for PD, MSA, DLB patients.
10. Subjects being treated with any anticoagulants or antiplatelet drugs, except aspirin at doses of 100 mg daily or lower within 2 weeks of the planned arterial cannula placement (if performed) for either the baseline or retest imaging.
11. Screening supine blood pressure > 150 mm Hg (systolic) or > 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure (BP) is > 150 mm Hg (systolic) or > 90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
12. Electrocardiographic (ECG) abnormalities of clinical significance as judged by the investigator. Screening supine 12-lead ECG demonstrating QTc > 450 msec at Screening.
13. Any contraindications to obtaining a brain MRI (except for Part 4 subjects), DaT-SPECT (except for Part 4 subjects) or PET (e.g., claustrophobia unresponsive to reassurance or low dose of an anxiolytic agent, metal implants not compatible with MRI or known hypersensitivity to the active substance or to any of the excipients) and ability to tolerate lying in the scanner for up to ~180 minutes.
14. Previous exposure to radiation for medical, scientific or other reasons which could have a high negative impact on the research subject, as judged by the investigator.
15. Treatment with any other investigational therapy within 5 drug elimination half-lives or 30 days (whichever is longer) prior to inclusion in the study.

    Additional Exclusion Criteria for Healthy Volunteers:
16. Current use of CNS active drugs, including antidepressant or neuroleptic medications is not permitted, anti-inflammatory drugs or sleep medications may be allowed at the discretion of the investigator.
17. History of neurological disease/condition that may interfere with the objectives of the study, as judged by the investigator.

    Additional Exclusion Criteria for Participants with α-synucleinopathy:
18. Medical history indicating a Parkinsonian syndrome other than idiopathic PD, including but not limited to, progressive supranuclear palsy, drug-induced parkinsonism, essential tremor, vascular parkinsonism, primary dystonia or corticobasal syndrome (CBS).
19. Known carriers of certain familial PD gene mutations (PRKN, PINK1, DJ1, LRRK2), based on previous source documentation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) assessed by severity (mild, moderate, severe, life threatening, death) and causal relationship (not related, unlikely related, possibly related or related) | From Informed Consent Signature (screening) to safety phone call after PET scan (i.e. up to 14 weeks in total)
Number of participants with clinically significant changes in vital signs measurements | During PET scan visit (i.e. at Day 0): before [18F]ACI-15916 injection and after the PET scan is completed
  Vital signs measurements will be performed after the PET scan is completed and will be compared with measurements performed before the injection of [18F]ACI-15916
Brain uptake of the tracer [18F]ACI-15916 | At the time of the [18F]ACI-15916 PET scan (i.e. at Day 0): 0-93 minutes after injection
  [18F]ACI-15916 uptake in relevant regions of interest of the brain will be measured with PET scan and the mean of each group (participants with α-synucleinopathies and healthy volunteers) will be calculated

SECONDARY OUTCOMES:
Assessment of simplified methods to quantify brain uptake of the tracer [18F]ACI-15916 | At the time of the [18F]ACI-15916 PET scan (i.e. at Day 0): 0-93 minutes after injection
  Reference tissue models will be used to quantify the brain uptake of the tracer [18F]ACI-15916 using an appropriate reference region in the brain. The mean will be calculated for each group (healthy volunteers and α-synucleinopathies)
Variability of the tracer brain uptake between two [18F]ACI-15916 PET scans (test/retest) | From the first PET scan (i.e. Day 0) to the second PET scan (i.e. Day 30)
  The repeatability/reliability of the [18F]ACI-15916 brain uptake measures will be assessed by calculating the variability (percentage difference) of the tracer brain uptake between the first and the second [18F]ACI-15916 PET scan for each participant in study Part 3, and the mean will be calculated.
Radiation dosimetry after one [18F]ACI-15916 PET scan | At the time of the [18F]ACI-15916 PET scan (i.e. at Day 0): 0-6 hours after injection
  The radiation dose absorbed by relevant vital organs and the total effective dose will be measured for each participant of study Part 4, and the mean of scanned participants will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Varrone, Prof., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided